CLINICAL TRIAL: NCT03497546
Title: Supervised Exercise Following Bariatric Surgery in the Treatment of Severe/Morbid Obesity: a Randomized Controlled Trial
Brief Title: Exercise Following Bariatric Surgery for Severe/Morbid Obesity (EFIBAR)
Acronym: EFIBAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); Complejo Hospitalario Torrecárdenas (CHT), Almería, Spain (Unknown)
Responsible Party: Principal Investigator, Enrique García Artero, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEP2016-74926-R
Record Dates: First submitted 2018-03-07; First posted 2018-04-13 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate
Keywords: Morbid obesity; Exercise; Weight loss; Cardiometabolic risk; Bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Motor Activity; Weight Loss | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly assigned (1:1) sequentially, as they will be submitted to bariatric surgery, to one of the two following groups:
  CON - Usual care (following international guidelines) after bariatric surgery. EX - Usual care plus supervised exercise program.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators, study coordinators, outcome assessors, and clinical staff will be blinded to the group allocation.
  Participants and providers of the exercise delivery will not be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Usual care PLUS concurrent (aerobic and strength) supervised exercise program of 16 weeks (3 sessions/week, 60 min/session, progressively increasing in volume and intensity). The program will be conducted by certified Exercise Science professionals.
  Interventions: Other: Exercise
- Control (No Intervention): Usual care routinely delivered after bariatric surgery, based on national (Spanish) and international recommendations, focused on nutritional status monitoring and diet/physical activity counseling.

INTERVENTIONS:
Other: Exercise — Concurrent (aerobic and strength) supervised exercise program: the program comprises 3 sessions/week (60 min/session) of aerobic and strength exercises of progressive volume and intensity. The program will follow the Consensus on Exercise Reporting Template (CERT) guidelines.
  Other Names: Exercise training
  Arms: Exercise

SUMMARY:
Severe/morbid obesity is an international public health issue that importantly increases the risk of cardiovascular events and cardiovascular and all-cause mortality. Likewise, severe/morbid obesity increases the risk of illness, reduces quality of life, and raises health-care costs. Bariatric surgery is the election method for the treatment of severe/morbid obesity, resulting in significant weight loss and remission of comorbidities. However, a relatively large proportion of bariatric patients regain weight and continue to be at high risk for cardiovascular disease and premature mortality. A healthy lifestyle following bariatric surgery is essential for optimizing and maintaining weight loss. Observational studies suggest that physical activity following bariatric surgery might be associated with additional weight loss and more effective weigh loss maintenance over time. However, very little experimental evidence exists regarding the effects of supervised exercise on obesity-related outcomes in this specific population.

The aim of the EFIBAR (Ejercicio FÍsico tras cirugía BARiátrica) randomized controlled trial is to determine the effects of a 16-week supervised concurrent (aerobic and strength) exercise intervention program, on weight loss (primary outcome), body composition, cardiometabolic risk, physical fitness and quality of life (secondary outcomes) in patients with severe/morbid obesity following bariatric surgery.

According to the study aims the investigators pursue the following hypothesis: Supervised exercise will result in larger weight loss than control.

ELIGIBILITY:
Inclusion Criteria:

* To comply with local bariatric surgery criteria:

  1. Patients with BMI ≥ 40 kg/m2 (or 35 kg/m2 with comorbidities).
  2. Acceptable surgical risk (defined by the approval of anesthetist).
  3. Obesity maintained for over 5 years.
  4. Failure of previous treatments.
  5. To sign informed consent for surgical treatment.
* Not to present contraindications for supervised physical exercise.
* To reside in the city of Almeria (Spain) or willingness/predisposition to attend the training sessions 3 times a week during 16 weeks

Exclusion Criteria:

* Severe psychiatric or neurological disorders such as schizophrenia, epilepsia, Alzheimer, Parkinson, personality disorders, eating behaviour disorders, untreated depression or suicidal tendencies.
* Adrenal or thyroid pathology that might cause obesity.
* Uncontrolled addiction to alcohol or drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Percent total weight loss (%TWL) [Biospace Co., InBody 270, USA] | Changes from baseline to 4-month and 1-year follow-up
  %TWL = [(pre-surgery weight - post-surgery weight) / (pre-surgery weight)] x 100

SECONDARY OUTCOMES:
Body composition: body fat | Changes from baseline to 4-month and 1-year follow-up
  Percent body fat (%) assessed by bioimpedance analysis (InBody 270, Biospace Co., USA)
Body composition: fat-free mass | Changes from baseline to 4-month and 1-year follow-up
  Fat-free mass (kg) assessed by bioimpedance analysis (InBody 270, Biospace Co., USA)
Body composition: fat-free mass index | Changes from baseline to 4-month and 1-year follow-up
  Fat-free mass index (kg/m2) assessed by bioimpedance analysis (InBody 270, Biospace Co., USA)
Body composition: central body fat | Changes from baseline to 4-month and 1-year follow-up
  Waist and hip circumferences (measured in cm with an anthropometric tape), waist / height ratio
Lipid profile assessed from blood sample | Changes from baseline to 4-month and 1-year follow-up
  Total cholesterol (mg/dl), HDL-cholesterol (mg/dl), LDL-cholesterol (mg/dl) and triglycerides (mg/dl)
Blood markers of glucose metabolism: glucose | Changes from baseline to 4-month and 1-year follow-up
  Glucose (mg/dL)
Blood markers of glucose metabolism: insulin | Changes from baseline to 4-month and 1-year follow-up
  Insulin (μUI/mL)
Blood markers of glucose metabolism: HOMA-IR | Changes from baseline to 4-month and 1-year follow-up
  Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Blood markers of glucose metabolism: glycated hemoglobin HbA1c | Changes from baseline to 4-month and 1-year follow-up
  Glycated hemoglobin HbA1c (%)
Brachial and central blood pressures (mmHg) | Changes from baseline to 4-month and 1-year follow-up
  Systolic and diastolic blood pressures assessed by Mobil-O-Graph
Arterial stiffness | Changes from baseline to 4-month and 1-year follow-up
  Pulse wave velocity (PWV, m/s) by Mobil-O-Graph
Plasma concentrations of inflammatory markers | Changes from baseline to 4-month and 1-year follow-up
  High-sensitivity C-reactive protein (hs-CRP)
Plasma concentrations of inflammatory markers | Changes from baseline to 4-month and 1-year follow-up
  Tumor necrosis factor (TNF-alpha)
Plasma concentrations of inflammatory markers | Changes from baseline to 4-month and 1-year follow-up
  Interleukin 6 (IL-6)
Plasma concentrations of liver metabolism enzymes | Changes from baseline to 4-month and 1-year follow-up
  GGT (gamma-glutamyltransferase)
Plasma concentrations of liver metabolism enzymes | Changes from baseline to 4-month and 1-year follow-up
  GPT (glutamate-pyruvate transaminase)
Plasma concentrations of liver metabolism enzymes | Changes from baseline to 4-month and 1-year follow-up
  GOT (glutamate-oxalacetate transaminase)
Plasma levels of Vitamin D | Changes from baseline to 4-month and 1-year follow-up
  Concentrations of 25-hydroxyvitamin D (ng/mL)
Heart rate variability (HRV) | Changes from baseline to 4-month and 1-year follow-up
  Assessed by heart rate monitor (Polar V800)
Health-related physical fitness: cardiorespiratory fitness | Changes from baseline to 4-month and and 1-year follow-up
  Cardiorespiratory fitness, assessed using a maximal treadmill test
Health-related physical fitness: upper body muscular strength | Changes from baseline to 4-month and and 1-year follow-up
  Upper body muscular strength, assessed using handgrip dynamometry (kg)
Health-related physical fitness: lower body muscular strength | Changes from baseline to 4-month and and 1-year follow-up
  Lower body muscular strength, assessed using the 30-seconds chair-stand test (number of repetitions)
Health-related physical fitness: upper body flexibility | Changes from baseline to 4-month and and 1-year follow-up
  Upper body flexibility, assessed using the back scratch test (cm)
Objectively-measured physical activity | Changes from baseline to 4-month and 1-year follow-up
  Assessed by accelerometry (ActiGraph, software ActiLife)
Health-Related Quality of Life (HRQoL): SF-36 | Changes from baseline to 4-month and 1-year follow-up
  Measured by the 36-item Short Form Health Survey (SF-36)
Health-Related Quality of Life (HRQoL): EQ-5D-3L | Changes from baseline to 4-month and 1-year follow-up
  Measured by European Quality of Life - 5 Dimensions-3Levels (EQ-5D-3L)
Symptomatology and function of hip / knee osteoarthritis: Pain | Changes from baseline to 4-month and 1-year follow-up
  Measured by the WOMAC (Western Ontario and McMaster Universities) Osteoarthritis Index. The PAIN scale within the WOMAC questionnaire contains 5 items, each one scoring from 0 (Nothing) to 4 (Very much), what makes a total score ranging from 0 (better) to 20 (worse).
Symptomatology and function of hip / knee osteoarthritis: Function | Changes from baseline to 4-month and 1-year follow-up
  Measured by the WOMAC (Western Ontario and McMaster Universities) Osteoarthritis Index. The FUNCTION scale within the WOMAC questionnaire contains 17 items, each one scoring from 0 (No trouble) to 4 (Very much difficult), what makes a total score ranging from 0 (better) to 68 (worse).
Symptomatology and function of hip / knee osteoarthritis: Stiffness | Changes from baseline to 4-month and 1-year follow-up
  Measured by the WOMAC (Western Ontario and McMaster Universities) Osteoarthritis Index. The STIFFNESS scale within the WOMAC questionnaire contains 2 items, each one scoring from 0 (Nothing) to 4 (Very much), what makes a total score ranging from 0 (better) to 8 (worse).
Depression, anxiety and stress | Changes from baseline to 4-month and 1-year follow-up
  Measured by the Depression, Anxiety and Stress Scale short form (DASS-21). The DASS-21 comprises three sub-scales assessing specific psychiatric symptoms (i.e., depression, anxiety, and stress). Each of these symptoms is assessed using seven items rated on a 4-point Likert-type scale (i.e., 0 = ''Did not apply to me at all''; 3 = ''Applied to me very much, or most of the time''). Summed score for each psychiatric symptom ranges from 0 to 21. Higher scores in each sub-scale indicate higher levels of depressive, anxiety or stress symptomatology. According to the specific nature of the three psychiatric symptoms assessed by the DASS-21, these are treated independently so that no total score is available.
Emotional, psychological and social well-being | Changes from baseline to 4-month and 1-year follow-up
  Measured by the Mental Health Continuum-Short Form (MHC-SF)
Cost-effectiveness analysis (CEA) | From baseline to 1-year follow-up
  The costs will consider those related to the surgery, the exercise program, prescription medication, sick leave, post-surgery complications and readmission rates, time and effort requiring each treatment, as well as possible dietary and informal care costs. Effectiveness will be considered as changes observed in the main clinical outcomes: weight loss and cardiometabolic risk (remission/relapse of hypertension, dyslipidemia and type 2 diabetes).
Cost-utility analysis (CUA) | From baseline to 1-year follow-up
  The costs will consider those related to the surgery, the exercise program, prescription medication, sick leave, post-surgery complications and readmission rates, time and effort requiring each treatment, as well as possible dietary and informal care costs. Utility will evaluate variation in quality of life experienced by participants, computed as changes in quality-adjusted life years (QALY) using SF-36 questionnaire.
Cost-utility analysis (CUA) | From baseline to 1-year follow-up
  The costs will consider those related to the surgery, the exercise program, prescription medication, sick leave, post-surgery complications and readmission rates, time and effort requiring each treatment, as well as possible dietary and informal care costs. Utility will evaluate variation in quality of life experienced by participants, computed as changes in quality-adjusted life years (QALY) using EQ-5D-3L questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique G Artero, Ph.D., Principal Investigator — Universidad de Almeria
Locations (1):
- Complejo Hospitalario Torrecárdenas (CHT), Almería, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be shared once the study is finalised and the main results are published. IPD can be obtained by contacting the responsible party (artero@ual.es).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Two years (24 months) after the study completion.
Access Criteria: The PI must be contacted and a minimum number of co-authors from the research team must be included in any publication.

REFERENCES:
- [Background] Villa-Gonzalez E, Barranco-Ruiz Y, Rodriguez-Perez MA, Carretero-Ruiz A, Garcia-Martinez JM, Hernandez-Martinez A, Torrente-Sanchez MJ, Ferrer-Marquez M, Soriano-Maldonado A, Artero EG; EFIBAR Study Group. Supervised exercise following bariatric surgery in morbid obese adults: CERT-based exercise study protocol of the EFIBAR randomised controlled trial. BMC Surg. 2019 Sep 5;19(1):127. doi: 10.1186/s12893-019-0566-9. PMID 31488115
- [Background] Artero EG, Ferrez-Marquez M, Torrente-Sanchez MJ, Martinez-Rosales E, Carretero-Ruiz A, Hernandez-Martinez A, Lopez-Sanchez L, Esteban-Simon A, Romero Del Rey A, Alcaraz-Ibanez M, Rodriguez-Perez MA, Villa-Gonzalez E, Barranco-Ruiz Y, Martinez-Forte S, Castillo C, Gomez Navarro C, Aceituno Cubero J, Reyes Parrilla R, Aparicio Gomez JA, Femia P, Fernandez-Alonso AM, Soriano-Maldonado A. Supervised Exercise Immediately After Bariatric Surgery: the Study Protocol of the EFIBAR Randomized Controlled Trial. Obes Surg. 2021 Oct;31(10):4227-4235. doi: 10.1007/s11695-021-05559-8. Epub 2021 Jul 15. PMID 34268680
- [Derived] Amaro Santos C, Cinza AM, Laranjeira A, Amaro M, Carvalho M, Martins S, Bravo J, Raimundo A. The impact of exercise on prevention of sarcopenia after bariatric surgery: The study protocol of the EXPOBAR randomized controlled trial. Contemp Clin Trials Commun. 2022 Dec 5;31:101048. doi: 10.1016/j.conctc.2022.101048. eCollection 2023 Feb. PMID 36568444
- See also: Study Protocol of the EFIBAR Randomized Controlled Trial — https://link.springer.com/article/10.1007/s11695-021-05559-8
- See also: CERT-based exercise study protocol of the EFIBAR randomised controlled trial — https://bmcsurg.biomedcentral.com/articles/10.1186/s12893-019-0566-9